CLINICAL TRIAL: NCT00428025
Title: Diclofenac for the Prevention of Post-ERCP Pancreatitis in Higher Risk Patients: A Prospective, Randomized, Double Blind, Placebo Controlled Trial.
Brief Title: Diclofenac for the Prevention of Post-ERCP Pancreatitis in Higher Risk Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: diclofenac trial hookey
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatitis
Keywords: pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo suppository (Placebo Comparator)
  Interventions: Drug: placebo
- diclofenac suppository (Active Comparator)
  Interventions: Drug: diclofenac

INTERVENTIONS:
Drug: diclofenac — 100 mg diclofenac rectal suppository
  Arms: diclofenac suppository
Drug: placebo — similar shape and size suppository
  Arms: placebo suppository

SUMMARY:
Inflammation of the pancreas (pancreatitis) is an uncommon but potentially serious complication of endoscopic retrograde cholangiopancreatography (ERCP), a specialized endoscopic examination of the ducts draining the liver and pancreas. Although many different strategies have been tried and studied in attempts to reduce this risk, few have been shown to make a significant difference. Those that have are either very expensive, difficult to administer, or both.

Diclofenac, an anti-inflammatory medication most often used to treat arthritis, has shown potential to decrease the risk of post-ERCP pancreatitis. It can be given after the procedure to patients at most risk for the complication, and has few side effects. This study will randomize people in the study to placebo or active medication, to determine if Diclofenac reduces the incidence of pancreatitis.

DETAILED DESCRIPTION:
Hypothesis:

Diclofenac, when administered immediately post ERCP in patients at higher risk of developing post-ERCP pancreatitis, will significantly reduce the incidence of this complication.

Intervention:

All patients undergoing ERCP not having exclusion criteria will be approached for participation prior to the procedure. At the end of the procedure, prior to transfer from the endoscopy suite, within 15 minutes of the end of the procedure, if the patient meets inclusion criteria, a study suppository will be administered.

The suppositories will be prepared by a study pharmacist according to a randomization list prepared by an independent biostatistician. They will be randomized using a permuted block design, in blocks of 20. The placebo is inert, and identical to the study medication, a 100 mg diclofenac rectal suppository. The code will not be broken until enrolment of patients is complete.

Patients, endoscopists, nurses, and the principal investigator will all be blinded to the randomization code.

Outcomes:

Post-ERCP acute pancreatitis is the primary outcome. Consensus definition of this is new typical (epigastric/retroperitoneal) pain combined with an elevation of serum lipase or amylase >3 times the upper limit of normal. Pain will be assessed through history and physical exam by an attending gastroenterologist the morning after the procedure, with documentation in the chart and research form of the presence or absence of pain. Serum amylase will be measured the morning after the procedure, between 7 and 10 am (approximately 18 hours post procedure). Most patients will be inpatients but outpatients will be included if they can be assessed through clinical exam and blood chemistry analysis the following morning. Patients will be contacted one week after the procedure to ensure no episode of abdominal pain or bleeding has been missed.

Statistics and Power Calculation

A two sided Fisher's Exact Test will be used to compare the proportion of patients developing post-ERCP pancreatitis in each group (placebo vs. active drug).

In the population selected, the estimated risk of pancreatitis is 15%. To demonstrate a decrease to 5%, 141 patients will be required in each group, with 80% power and an alpha error 0.05. Secondary outcomes will include severity of pancreatitis, hyperamylasemia, length of stay, and mortality. Safety data regarding renal function and GI bleeding will also be collected.

ELIGIBILITY:
Inclusion Criteria:

These were chosen based on a review of the major studies evaluating risk factors for post-ERCP pancreatitis. Any of the following factors placing a patient at high risk (>10%) of post ERCP pancreatitis:

* Patient characteristics: Prior history of post-ERCP pancreatitis, prior history of acute pancreatitis, suspected Sphincter of Oddi dysfunction, or normal bilirubin;
* Procedure related factors: Moderate (6-15 attempts) and difficult (>15 attempts) bile duct cannulation, balloon dilation of the biliary sphincter, pre-cut papillotomy, pancreatic sphincterotomy.

Exclusion Criteria:

* Ongoing acute or chronic pancreatitis;
* Previous biliary sphincterotomy;
* Contra-indications to non-steroidal anti-inflammatory medications (allergy, reduced renal function, recent upper gastrointestinal bleeding);
* Ingestion of an NSAID ( nonsteroidal anti-inflammatory drug) in the previous 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
post-ercp pancreatitis | 24 hours

SECONDARY OUTCOMES:
severity of pancreatitis, side effects | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada